## **Informed consent form**

## **Subjects informed consent statement:**

- 1, I have read the informed consent and fully understood all the content.
- 2, I have the opportunity to ask questions and all the questions have been answered.
- 3, I understand that participating in this study is voluntary.
- 4, I can choose not to participate in this study, and my medical treatment, rights and interests will not be affected.
- 5, If I need any other treatment, or I don't follow the research plan, or I have something to do with the study for injury or any other reasons, the researchers may terminate my participation in this study.

| terminate my participation in this study. | 0110, 0110 1 00001 011010 11101 |
|---|---|
| 6, I will receive a copy of the signed "informed consent form" | '' . |
| Signature: | |
| Date: | |
| Researchers informed consent statement: | |
| 1, I have informed the subjects or their representatives of procedures, risks and benefits of the study. | f the purposes, methods, |
| 2, Given them enough time to read the informed conser-<br>questions. | nt, and I answer all the |
| 3, I have informed the subjects of the contact information who 4, I have informed the subjects or their legal representatives the withdraw from this study during the period at any time. | - |
| Signature: | |
| Date: | |